CLINICAL TRIAL: NCT01614444
Title: Using Complementary and Alternative Medicine (CAM) to Promote Stress Resilience in Those With Co-Occurring Mild TBI and PTSD
Brief Title: Acupressure and Stress Resilience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Collaborators: University of Colorado, Boulder (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lisa Brenner, Director of MIRECC (Mental Illness Research, Education and Clinical Center, VA Eastern Colorado Health Care System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COMIRB# 12-0452
Record Dates: First submitted 2012-06-05; First posted 2012-06-08 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Post-traumatic Stress Disorder (PTSD); Mild Traumatic Brain Injury (mTBI)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Concussion

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Acupressure Treatment (Active Comparator)
  Interventions: Other: Active Acupressure Treatment
- Placebo Acupressure Treatment (Placebo Comparator)
  Interventions: Other: Placebo Acupressure Treatment

INTERVENTIONS:
Other: Active Acupressure Treatment — Participant will receive 8 active acupressure treatments.
  Arms: Acupressure Treatment
Other: Placebo Acupressure Treatment — Participants will receive 8 placebo acupressure treatments.
  Arms: Placebo Acupressure Treatment

SUMMARY:
The current study will assess the efficacy of acupressure, a type of complementary and alternative medicine (CAM) in the Veteran population. Veterans with co-occurring mild traumatic brain injury (mTBI) and post-traumatic stress disorder (PTSD) will be consented and randomly assigned to either an active or placebo acupressure treatment series of 8 sessions. The investigators will determine if acupressure affects aspects of day-to-day function, such as memory, sleep, mood, psychiatric health and stress resilience. This information will help identify potential treatment strategies to improve quality of life and overall function in this particular Veteran population.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-60
* Diagnosis of mild TBI and PTSD as assessed by interview and/or chart review
* Currently receiving or eligible to receive physical and/or mental healthcare through the VA Eastern Colorado Health Care System

Exclusion Criteria:

* History of other significant neurological disease (e.g., Alzheimer's, Parkinson's, multiple sclerosis etc.) as assessed by interview and/or chart review. Such conditions could affect outcome measures independently, thereby creating an experimental confound.
* History or diagnosis of lifetime moderate to severe TBI, as assessed by interview and/or chart review.
* History of psychotic disorder or bipolar I disorder as assessed by structured interview. Such conditions could affect outcome measures independently, thereby creating an experimental confound.
* Inability to read the informed consent document or adequately respond to questions regarding the informed consent procedure.
* Prior experience with acupressure, as this would result in individuals potentially being able to detect Placebo treatments if randomly assigned to that group.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-06-13 (Actual); Primary Completion 2014-08-11 (Actual); Study Completion 2017-03-07 (Actual)

PRIMARY OUTCOMES:
Trier Social Stress Test | 72 hours post final acupressure treatment

CONTACTS AND LOCATIONS:
Overall Officials: Theresa D Hernandez, Ph.D., Principal Investigator — Senior Investigator and Research Psychologist Eastern Colorado Healthcare System, VISN19, MIRECC; Lisa A Brenner, Ph.D., Principal Investigator — Eastern Colorado Healthcare System VISN 19 MIRECC Director
Locations (1):
- Denver VAMC, Denver, Colorado, United States